CLINICAL TRIAL: NCT06952088
Title: Face Mask vs Laryngeal Mask in Neonatal Resuscitation: A Study on Manikins
Brief Title: Face Mask vs Laryngeal Mask in Neonatal Resuscitation
Acronym: ManiMask2025
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 7557
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Neonatal Complication; Neonatal Asphyxia
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- health care Workers (Other): Healthcare Workers (physicians, nurses and midwives) of Neonatal Unit and Delivery Room of Fondazione Policlinico Gemelli Hospital IRCCS
  Interventions: Other: Training on Neonatal Resuscitation

INTERVENTIONS:
Other: Training on Neonatal Resuscitation — Improve training of health care personnel (physicians, nurses and midwives) on neonatal resuscitation through manikin simulation using two different devices: a face mask and a laryngeal mask. Before the simulations begin, each participant will receive a brief introduction on the technical characteristics of the manikin and how to use the two masks. A stopwatch will be used to record the time required to achieve effective ventilation, defined by the expansion of one-third of the newborn manikin's rib cage. Consideration will also be given to whether corrective maneuvers will need to be performed during the use of each mask and the timing with which these maneuvers will be applied. Finally, a pseudonymous questionnaire will be administered to participants to assess their perceptions of the ease of use of each mask.

SUMMARY:
The goal of this single-centre interventional study without medication neither device (for procedure) is to improve training of health care personnel (physicians, nurses, and midwives) on neonatal resuscitation through manikin simulation.

The main questions it aims to answer are:

* Is it possible to compare the ease of use and speed of application of the laryngeal mask versus the face mask in ventilating the newborn during simulated manikin training?
* What are the differences in the time required to achieve optimal skills in using the two masks?
* What is health care personnel's level of confidence in using laryngeal mask versus face mask?

DETAILED DESCRIPTION:
Maintaining airways and ensuring effective ventilation are the primary goals in the neonatal resuscitation algorithm.To achieve it, there are several devices, more or less invasive, such as a face mask, laryngeal Mask or tracheal tube.Among these, Laryngeal Mask can have significant advantages, including ease of use and speed of application even if used by inexperienced health personnel after a short training program.

The protocol involves the use of a neonatal manikin, which is already in the use at our simulation center. Ventilation of the manikin will be conducted using two possible masks: a face mask and a laryngeal mask. Before the simulations begin, each participant will receive a brief introduction on the technical characteristics of the manikin and how to use the two masks. A stopwatch will be used to record the time required to achieve effective ventilation, defined by the expansion of one-third of the newborn manikin's rib cage. Consideration will also be given to whether corrective maneuvers will need to be performed during the use of each mask and the timing with which these maneuvers will be applied.

Finally, a pseudonymous questionnaire will be administered to participants to assess their perceptions of the ease of use of each mask.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare Workers (physicians, nurses, and midwives) of the Neonatal Unit and Delivery Room of Fondazione Policlinico Gemelli Hospital IRCCS Rome
* Signature of an informed consent

Exclusion Criteria:

* Healthcare Workers (physicians, nurses, and midwives) NOT of the Neonatal Unit and Delivery Room of Fondazione Policlinico Gemelli Hospital IRCCS Rome
* Failure to sign up for informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of ease of use and speed of application of the laryngeal mask versus the face mask in ventilating the newborn during simulated manikin training | During Training session
  . A stopwatch will be used to record the time required to achieve effective ventilation, defined by the expansion of one-third of the newborn manikin's rib cage.

SECONDARY OUTCOMES:
Comparison of differences in the time required to achieve optimal skills in using the two masks | During Training session
  . A stopwatch will be used to record the time required to achieve effective ventilation, defined by the expansion of one-third of the newborn manikin's rib cage.
Evaluation of health care personnel's level of confidence in using laryngeal mask versus face mask | During Training session
  A pseudonymous questionnaire will be administered to participants to assess their perceptions of the ease of use of each mask

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Priolo, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS; UOC Neonatologia
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS; UOC Neonatologia, Roma, Italy